CLINICAL TRIAL: NCT00068315
Title: A Phase I Trial of PS-341 and Fludarabine for Relapsed and Refractory Indolent Non-Hodgkin's Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: Bortezomib and Fludarabine With or Without Rituximab in Treating Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00044; NCI-2009-00044 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ICC 3402; CDR0000321394; ICC 3402 (Other: Case Western Reserve University); 6126 (Other: CTEP); U01CA062502 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hematopoietic/Lymphoid Cancer; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Bortezomib; fludarabine phosphate; Rituximab

ARMS (1):
- Treatment (bortezomib, fludarabine, rituximab) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and fludarabine IV over 30 minutes on days 1-3 or 1-5. Patients may also receive rituximab IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: bortezomib; Drug: fludarabine phosphate; Biological: rituximab

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan

SUMMARY:
This phase I trial is studying the side effects and best dose of bortezomib when given together with fludarabine with or without rituximab in treating patients with relapsed or refractory indolent non-Hodgkin's lymphoma or chronic lymphocytic leukemia. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy, such as fludarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with fludarabine with or without rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and toxicity of bortezomib and fludarabine with or without rituximab in patients with relapsed or refractory indolent non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

II. Determine the maximum tolerated dose of bortezomib in combination with fludarabine in these patients.

III. Determine the biological effect of this regimen on apoptotic markers, cell cycle kinase inhibitors, and DNA repair in these patients.

OUTLINE: This is a multicenter, dose-escalation study of bortezomib.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and fludarabine IV over 30 minutes on days 1-3 or 1-5. Patients may also receive rituximab IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL) OR indolent non-Hodgkin's lymphoma (NHL) of any of the following subtypes:

  * Follicular lymphoma:

    * Grade I follicular small cleaved cell;
    * Grade II follicular mixed cell;
    * Grade II follicular large cell;
    * Diffuse small cleaved cell;
    * Small lymphocytic lymphoma;
    * Lymphoplasmacytic lymphoma (Waldenstrom's macroglobulinemia)
* AND

  * Extranodal marginal zone B-cell lymphoma (mucosa-associated lymphoid tissue [MALT] lymphoma);
  * Nodal marginal zone B-cell lymphoma (monocytoid B-cell lymphoma);
  * Splenic marginal zone lymphoma (splenic lymphoma with villous lymphocytes);
  * Mantle cell lymphoma:

    * No blastic phase mantle cell lymphoma
* Relapsed or refractory, progressive disease:

  * First, second, or third relapse
* Measurable disease, meeting 1 of the following criteria:

  * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan (for NHL patients);
* OR:

  * Lymphocytosis > 50,000/mm3 OR evidence of progressive bone marrow infiltration failure (e.g., hemoglobin 10 g/dL) OR thrombocytopenia (i.e., platelet count < 100,000/mm3) with > 30% infiltration of bone marrow by leukemia (for CLL patients)
* No measurable lymphadenopathy (for CLL and Waldenstrom's macroglobulinemia patients)
* No evidence of CNS lymphoma
* Performance status:

  * ECOG 0-2
* Life expectancy:

  * More than 12 weeks
* No history of uncontrolled orthostatic hypotension
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No uncontrolled concurrent illness
* No grade 2 or greater neuropathy
* No history of allergy or anaphylaxis to mannitol, bortezomib, fludarabine, or boron
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* At least 4 weeks since prior monoclonal antibody (MoAB) therapy:

  * Patients who have received MoAB therapy within the past 3 months must have documented disease progression since receiving this therapy
* No prior allogeneic stem cell transplantation
* More than 4 weeks since prior chemotherapy
* Prior fludarabine allowed
* At least 1 week since prior steroids
* At least 3 months since prior radio-immunotherapy
* More than 4 weeks since prior radiotherapy
* No prior bortezomib
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 75,000/mm3 (greater than 50,000/mm3 if lymphomatous bone marrow involvement is present)
* Bilirubin no greater than 2.0 mg/dL
* AST/ALT no greater than 4 times normal
* Creatinine clearance greater than 40 mL/min
* No other concurrent investigational agents or treatments for the malignancy
* No brain metastases
* OR:

Quantitation of IgM paraprotein (for Waldenstrom's macroglobulinemia patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-07; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) assessed by Common Toxicity Criteria version 2.0 | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Cooper, Principal Investigator — Case Western Reserve University
Locations (7):
- United States (7):
  - Mercy Medical Center, Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Seidman Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - University Suburban Medical Center, South Euclid, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio